CLINICAL TRIAL: NCT03234452
Title: Evaluation of the Beneficial Effects of a Probiotic Product (Lactoflorene Plus) in Healthy Adult Subjects in Particular Psychological Stress Conditions.
Brief Title: Evaluation of the Beneficial Effects of a Probiotic Product in Healthy Adult Subjects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefarmaco OTC SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Lactoflorene plus
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Disbiosis; Abdominal Pain; Constipation; Diarrhea; Stress
Keywords: Lactoflorene plus; Bifidobacterium animalis subsp. lactis, BB-12®; Lactobacillus acidophilus, LA-5®; Lactobacillus paracasei subsp. paracasei, L. CASEI 431®; Inflammation; gut permeability; disbiosis; probiotic; IgA; IL10
MeSH Terms: conditions — Dysbiosis; Abdominal Pain; Constipation; Diarrhea; Inflammation

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled, cross-over trial performed at one centre
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactoflorene plus (Experimental): 10 ml mixture of Lactobacillus acidophilus LA-5®, Bifidobacterium animalis subsp. lactis, BB-12®, Lactobacillus paracasei subsp. paracasei, L. CASEI 431® , Bacillus coagulans BC513, zinc and B-vitamins (niacin, B1, B2, B5, B6, B12 and folic acid) twice a day
  Interventions: Dietary Supplement: Lactoflorene plus
- Placebo Lactoflorene plus (Placebo Comparator): Identical placebo mixture without probiotics, B-vitamins and zinc. The active and placebo products had similar appearance, taste and smell and were provided in identical bottles of 10 ml with identical labelling.
  Interventions: Dietary Supplement: Placebo Lactoflorene plus

INTERVENTIONS:
Dietary Supplement: Lactoflorene plus — 2 vials with dosing cap (10 mL) a day per os
  Arms: Lactoflorene plus
Dietary Supplement: Placebo Lactoflorene plus — 2 vials with dosing cap (10 mL) a day per os
  Arms: Placebo Lactoflorene plus

SUMMARY:
A randomized, double-blind, placebo-controlled, cross-over trial performed at one centre in Italy to explore the ability of a multistrain probiotic mixture, to modulate markers of inflammation and intestinal barrier function and gastrointestinal symptoms in healthy volunteers with self-reported anxiety.

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects were healthy men and women, 20-35 years old, with a STAI scale, form Y, module 1 (state anxiety) score of ≥ 35 and ≥40, for men and women, respectively.

Exclusion Criteria:

Most important exclusion criteria were history or diagnosis of GI disease, oral antibiotics within 30 days prior to the screening visit, and use of drugs, food or herbal supplements for digestive symptoms.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2016-07-21 (Actual); Study Completion 2017-04-18 (Actual)

PRIMARY OUTCOMES:
NK activity | 45 days
  Verify that Natural Killer activities concentration is significantly higher in the experimental Group compared to the placebo group

SECONDARY OUTCOMES:
IgA, IL8, TNF-Alpha, IL10 | 45 days
Cortisol, alpha-amylase , chromogranin A | 45 days
microbiota composition investigation | 45 days
Gastrointestinal symptoms (abdominal pain, aerophagia, diarrhea, constipation, diarrhea/constipation alternation ) | 45 days

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Ricerche Cliniche di Verona Srl,, Verona, (Vr), Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soldi S, Tagliacarne SC, Valsecchi C, Perna S, Rondanelli M, Ziviani L, Milleri S, Annoni A, Castellazzi A. Effect of a multistrain probiotic (Lactoflorene(R) Plus) on inflammatory parameters and microbiota composition in subjects with stress-related symptoms. Neurobiol Stress. 2018 Nov 7;10:100138. doi: 10.1016/j.ynstr.2018.11.001. eCollection 2019 Feb. PMID 30937345